CLINICAL TRIAL: NCT07099326
Title: Examining the Effects of Interactive Versus Conventional Video-Based Education on Activation, Treatment Adherence, and Weight Changes in Dialysis Patients: A Randomized Clinical Trial Protocol
Brief Title: Interactive vs. Standard Video Education for Improving Outcomes in Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sogand Sarmadi, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IR.SBMU.PHARMACY.REC.1404.067
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis; Nurse; Educational Videos; Patient Activation; Weight Change; Treatment Adherence
Keywords: Interactive Video-Based Education; Conventional Video-Based Education; Patient Activation; Patient Treatment Adherence; Patients' Weight Changes; Dialysis
MeSH Terms: conditions — Patient Participation; Body Weight Changes; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive Video-Based Intervention (Experimental): Participants in this arm will undergo a two-phase educational intervention with a total duration of six hours. In the first phase, patients will access an interactive video series on end-stage renal disease (ESRD) and its treatment options via an online platform. The series consists of ten 30-minute sessions delivered daily. The videos include interactive elements such as pop-up questions and multiple-choice assessments, with responses monitored by an instructor. All participants will receive prior training on how to use the system. In the second phase, patients will attend a one-hour instructor-led group discussion to review and consolidate key concepts.
  Interventions: Other: Educational Method Using Interactive Video
- Conventional Video-Based Education (Experimental): Participants in this arm will receive a two-phase educational intervention lasting a total of six hours. In the first phase, patients will access a series of conventional (non-interactive) educational videos on end-stage renal disease (ESRD) and treatment options via an online platform. The series consists of ten 30-minute sessions delivered daily. In the second phase, patients will participate in a one-hour instructor-led group discussion to review the video content, explore key concepts, and consolidate their understanding. Discussions will be facilitated by an experienced instructor familiar with the video content.
  Interventions: Other: Educational Method Using Conventional Video
- Control Group (Usual Care) (No Intervention): Participants in this group will receive the standard educational care provided at their respective centers. This typically includes nurse-delivered patient education, distribution of educational pamphlets, and follow-up by the unit's assigned nurse educator.

INTERVENTIONS:
Other: Educational Method Using Interactive Video — Phase 1 - Interactive Video-Based Training (10 sessions of 30 minutes each):
  Patients will access the platform via the website https://spotplayer.ir/ and watch a comprehensive interactive video related to end-stage renal disease (ESRD) and its replacement therapies. This video consists of ten 30-minute sessions, uploaded at the rate of one session per day. During the viewing, pop-up questions will appear, which patients are required to answer. Different response options will lead to the presentation of different educational scenarios. In addition, multiple-choice questions related to the content will be included throughout the video, and patients must record their answers in the system. The instructor will be able to review these responses through a management dashboard. It is worth noting that all patients will have previously received the necessary training to use the interactive videos, including Q&A sessions designed to ensure sufficient skill acquisition in utilizing the interact
  Arms: Interactive Video-Based Intervention
Other: Educational Method Using Conventional Video — This educational intervention will be carried out in two phases with a total duration of six hours. A total of 55 patients will participate in this study, organized into groups of five and guided by an experienced instructor familiar with the interactive video-based educational system.
  Phase 1 - Conventional Video-Based Training (10 sessions of 30 minutes each):
  Patients will access the platform through the website https://spotplayer.ir/ and watch in-depth educational videos related to end-stage renal disease (ESRD) and its replacement therapies. The video content consists of ten 30-minute sessions, which will be uploaded for the patients at the rate of one session per day.
  Phase 2 - Consolidation and Reinforcement Session (1 hour):
  After completing the ten video sessions, patients will participate in group discussions to analyze the scenarios, topics, and questions presented in the videos. The instructor will facilitate the discussions, summarize the outcomes, and assess the over
  Arms: Conventional Video-Based Education

SUMMARY:
The goal of this clinical trial is to find out if educational videos-especially interactive ones-can help people on dialysis better manage their treatment.

Researchers want to answer the following main questions:

Can interactive or conventional video-based education help patients better understand and follow their treatment plan? Does this type of education improve patients' ability to control their weight changes between dialysis sessions? Does this type of education improve patients' activation? Is interactive video education more effective than regular (non-interactive) video education?

What Will Happen in the Study:

Adults on hemodialysis will take part in the study.

They will be randomly assigned to one of three groups:

Group A: Will receive 10 interactive educational video sessions (30 minutes each).

Group B: Will receive the same videos but in a non-interactive format. Group C (Control Group): Will receive routine education normally given at the dialysis center.

Videos will be watched on a web platform. Interactive videos include pop-up questions and scenario-based feedback.

All participants will be followed up immediately, 1 month, and 3 months after the program ends.

What Participants Will Do:

Watch educational videos over several days (totaling 5 hours).

Answer questions and engage in follow-up group discussions.

Complete surveys about their knowledge, treatment adherence, and health behaviors.

Get weighed before and after dialysis sessions to monitor fluid retention.

This study aims to improve how dialysis patients manage their condition and to help healthcare providers design better educational tools.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in the study;
2. Literate (ability to read and write);
3. Alertness and orientation to time, place, and person sufficient to respond to questions;
4. No history of hearing or visual impairments;
5. No cognitive disorders;
6. Possession of a personal mobile phone or any other device capable of running interactive videos, and the ability to use it;
7. No use of psychoactive medications;
8. Confirmed diagnosis of chronic kidney disease by a nephrology specialist and having a medical record in the dialysis unit;
9. Age between 18 and 65 years.

Exclusion Criteria:

1. Withdrawal from the study at any stage;
2. Failure to receive and watch the provided videos;
3. Patient death;
4. Transfer to a healthcare center outside the coverage of Shahid Beheshti University of Medical Sciences.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
Patients Activation Measure | Baseline (prior to the intervention) Immediately after the completion of the intervention One month post-intervention Three months post-intervention
  Patient activation refers to an individual's knowledge, skills, confidence, and willingness to manage their own health and healthcare. In this study, patient activation is considered a primary behavioral outcome, as the educational intervention is designed to empower participants to take a more active role in managing their dialysis treatment and overall health. The Patient Activation Measure (PAM), developed by Hibbard and colleagues, consists of 13 items and is a valid and reliable tool for assessing patient activation in the field of nephrology. Responses are recorded using a five-point Likert scale ("Strongly disagree" = 1, "Disagree" = 2, "Agree" = 3, "Strongly agree" = 4, and "Not applicable" = no score). The raw total scores range from 13 to 52, with lower scores indicating lower activation levels and higher scores indicating higher activation levels (41).

SECONDARY OUTCOMES:
Treatment Adherence | Baseline (prior to the intervention) Immediately after the completion of the intervention One month post-intervention Three months post-intervention
  The End-Stage Renal Disease Adherence Questionnaire (ESRD-AQ) is a self-report instrument consisting of 46 items across five domains, designed to assess patient adherence to treatment in four areas: attendance at hemodialysis sessions, medication adherence, fluid restrictions, and dietary recommendations. The first section of the questionnaire collects general information about patients' knowledge of ESRD and their history of renal replacement therapy (5 items). The subsequent four sections assess adherence to hemodialysis attendance (14 items), medication use (9 items), fluid restriction (10 items), and dietary recommendations (8 items), respectively. Responses are recorded using a combination of Likert scales, multiple-choice questions, and yes/no formats. The total score ranges from 0 to 1200, with higher scores indicating greater adherence to treatment (43). The reliability of this instrument was confirmed by Rafiei et al. (2014), with a Cronbach's alpha of 0.91 and a test-retest
Patient Weight Changes | Baseline (prior to the intervention) Immediately after the completion of the intervention One month post-intervention Three months post-intervention
  In this study, interdialytic weight gain (IDWG) will be assessed by measuring patients' weight immediately before connection to the hemodialysis machine and immediately after the completion of each session, following a standardized protocol. All weight measurements will be conducted using a calibrated medical digital scale (calibrated monthly). Patients will consistently be weighed wearing a standardized light dialysis gown, after emptying their bladder and refraining from food or beverage intake. Additionally, all personal items (such as shoes, bags, and jewelry) will be removed prior to weighing. Trained staff or the researcher will carefully record all measurements at fixed time points (pre-dialysis and post-dialysis) to ensure data consistency and allow accurate comparison of weight changes throughout the treatment period.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sarmadi S, Sanaie N, Zare-Kaseb A. Comparing the effects of interactive and conventional video education on activation, treatment adherence, and weight changes in dialysis patients: A randomized clinical trial protocol. PLoS One. 2025 Oct 15;20(10):e0334498. doi: 10.1371/journal.pone.0334498. eCollection 2025. PMID 41091721